CLINICAL TRIAL: NCT04510090
Title: Randomized, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of EP547 in Healthy Subjects and Subjects With Cholestatic or Uremic Pruritus
Brief Title: Evaluate the Safety, Tolerability, and PK of EP547 in Healthy Subjects and Subjects With Cholestatic or Uremic Pruritus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Escient Pharmaceuticals, Inc (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP-547-101
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Pruritus; Cholestasis; Kidney Failure
MeSH Terms: conditions — Pruritus; Cholestasis; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EP547 Single Dose (Experimental): Single doses of EP547
  Interventions: Drug: EP547
- EP547 Multiple Doses (Experimental): Multiple doses of EP547
  Interventions: Drug: EP547
- Placebo Single Dose (Placebo Comparator): Single doses of placebo
  Interventions: Drug: Placebo
- Placebo Multiple Doses (Placebo Comparator): Multiple doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EP547 — EP547
  Arms: EP547 Multiple Doses; EP547 Single Dose
Drug: Placebo — Placebo
  Arms: Placebo Multiple Doses; Placebo Single Dose

SUMMARY:
This first in human, Phase 1/1b trial will evaluate the safety, tolerability, and pharmacokinetics of single and multiple ascending doses of EP547 in healthy subjects and subjects with cholestatic or uremic pruritus.

DETAILED DESCRIPTION:
This study consists of both single and multiple ascending doses in healthy subjects and in subjects with cholestatic or uremic pruritus.

Up to 48 healthy subjects will receive a single dose of EP547 or placebo. There will be a screening period of up to 28 days prior to the first dose, and a follow up visit 7 days after dosing is completed.

24 healthy subjects will receive multiple doses of EP547 or placebo for 7 days. There will be a screening period of up to 28 days prior to the first dose, and a follow up visit 7 days and then 14 days after dosing is completed.

6 subjects with cholestatic disease will receive a single dose of EP547. There will be a screening period of up to 28 days prior to the first dose, and a follow up visit 7 days after dosing is completed.

Up to 16 subjects with cholestatic pruritus will receive multiple doses of EP547 or placebo for 7 days. There will be a screening period of up to 28 days prior to the first dose, and a follow up visit 7 days and then 14 days after dosing is completed.

6 subjects with uremic disease will receive a single dose of EP547. There will be a screening period of up to 28 days prior to the first dose, and a follow up visit 7 days after dosing is completed.

Up to 16 subjects with uremic pruritus will receive multiple doses of EP547 or placebo for 7 days. There will be a screening period of up to 28 days prior to the first dose, and a follow up visit 7 days and then 14 days after dosing is completed.

12 healthy subjects will receive two doses of EP547 under fasted or fed condition.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects:

* Age 18 to 60 years, inclusive
* Body mass index greater than or equal to 19 to less than or equal to 35 kg/m2
* Medically healthy with no clinically significant medical history, physical examination, vital sign, standard 12- lead ECG, chemistry, hematology, urinalysis, or coagulation results at Screening as deemed by the Investigator
* Male and female subjects must use adequate birth control and agree not to donate sperm or eggs for the time periods specified in the protocol

Subjects with Cholestatic Pruritus:

* Age 18 to 80 years, inclusive
* Has a cholestatic disorder
* Has experienced daily or near-daily moderate to severe pruritus for greater than 4 weeks before Screening and at study entry has itch scores indicative of moderate to severe pruritus
* If currently taking medications to treat the cholestatic disorder, must be on a stable dose for greater than 12 weeks before Screening and plans to maintain the regimen throughout the study
* If currently taking medications known to impact pruritus, must be on a stable dose for greater than 4 weeks before Screening and plans to maintain the regimen throughout the study
* Male and female subjects must use adequate birth control and agree not to donate sperm or eggs for the time periods specified in the protocol

Subjects with Uremic Pruritus

* Age 18 to 80 years, inclusive
* Has ESRD and is receiving hemodialysis 3× per week
* Has experienced daily or near-daily moderate to severe pruritus for greater than 4 weeks before Screening and at study entry has itch scores indicative of moderate to severe pruritus
* If currently taking medications known to impact pruritus, must be on a stable dose for greater than 4 weeks before Screening and plans to maintain the regimen throughout the study
* Male and female subjects must use adequate birth control and agree not to donate sperm or eggs for the time periods specified in the protocol

Exclusion Criteria:

Healthy Subjects:

* Any prescription medications within 14 days of Screening
* Positive result for HIV HBV, or HCV at Screening
* History of malignancy within the past 5 years
* Tobacco product or electronic cigarette use within 90 days of Day -1
* Positive drug, alcohol, or cotinine screen results at Screening or Day -1
* Significant history of abuse of drugs, solvents, or alcohol in the past 2 years

Subjects with Cholestatic Pruritus:

* Scheduled to receive a liver transplant during the study (placement on a transplant waiting list is not exclusionary)
* Is receiving ongoing UVB treatment or anticipates receiving such treatment during the study
* Pruritus is secondary to biliary obstruction
* History or presence of hepatocellular carcinoma, hepatic abscess, or acute portal vein Thrombosis

Subjects with Uremic Pruritus:

* Scheduled to receive a kidney transplant during the study (placement on a transplant waiting list is not exclusionary)
* Is receiving ongoing UVB treatment or anticipates receiving such treatment during the study
* Known noncompliance with hemodialysis treatment that, in the opinion of the Investigator, would impede completion or validity of the study
* Pruritus is attributed mainly to any disease unrelated to kidney disease, is only present during the hemodialysis sessions, or is attributed to a skin disorder that occurs in this population with associated itch (eg, acquired perforating dermatosis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - CMAX Clinical Research, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Auckland Clinical Studies (ACS), Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted on 85 subjects at 4 sites in Australia and New Zealand. This study consisted of 7 segments: single ascending dose in healthy subjects (SAD-HS), multiple ascending dose in healthy subjects (MAD-HS), food effect in healthy subjects (FE-HS), single dose in subjects with cholestatic pruritus (SD-CP), multiple dose in subjects with cholestatic pruritus (MD-CP), single dose in subjects with uremic pruritus (SD-UP), and multiple dose in subjects with uremic pruritus (MD-UP).
Pre-assignment Details: A total of 89 subjects (85 unique subjects) participated in the study. SAD-HS n=40 MAD-HS n=24 FE-HS n=5 SD-CP n=5 SD-UP n=6 MD-CP n=3 MD-UP N=6 (4 subjects participated in both SD-UP and MD-UP)
Groups:
- Placebo: Participants in all segments received placebo matched to EP547.
- EP547 20 mg: Participants in MD-UP segment received 20 mg of EP547 QD for 7 days.
- EP547 25 mg: Participants in SAD-HS segment received a single 25 mg dose of EP547. Participants in MAD-HS segment received 25 mg of EP547 QD for 7 days.
- EP547 30 mg: Participants in MD-CP segment received 30 mg of EP547 QD for 7 days.
- EP547 75 mg: Participants in SAD-HS segment received a single 75 mg dose of EP547. Participants in MAD-HS segment received 75 mg of EP547 QD for 7 days. Participants in FE-HS segment received a single 75 mg dose of EP547 under fed or fasted condition, separated by a washout period.
  Participants in SD-CP and SD-UP segments received a single 75 mg dose of EP547.
- EP547 225 mg: Participants in SAD-HS segment received a single 225 mg dose of EP547. Participants in MAD-HS segment received 225 mg of EP547 QD for 7 days.
- EP547 450 mg: Participants in SAD-HS segment received a single 450 mg dose of EP547.
- EP547 675 mg: Participants in SAD-HS segment received a single 675 mg dose of EP547.
Period: SAD-HS
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Started | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6
Completed | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MAD-HS
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Started | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0
Completed | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: FE-HS
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Started | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: SD-CP
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Started | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SD-UP
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Started | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MD-CP
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Started | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MD-UP
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Started | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg | Total
Number analyzed (Participants) | 19 | 4 | 12 | 2 | 28 | 12 | 6 | 6 | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: This study consisted of 7 segments: 1) single ascending dose in healthy subjects (SAD-HS), 2) multiple ascending dose in healthy subjects (MAD-HS), 3) food effect in healthy subjects (FE-HS), 4) single dose in subjects with cholestatic pruritus (SD-CP), 5) multiple dose in subjects with cholestatic pruritus (MD-CP), 6) single dose in subjects with uremic pruritus (SD-UP), and 7) multiple dose in subjects with uremic pruritus (MD-UP).
  Years
    SAD-HS: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS | 27.3 (9.9) |  | 30.7 (12.3) |  | 32.5 (9.1) | 32.7 (11.1) | 30.2 (4.2) | 36.2 (4.2) | 31.2 (9.36)
    MAD-HS: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS | 32.8 (12.2) |  | 30.0 (13.5) |  | 42.0 (14.1) | 36.3 (16.3) |  |  | 35.3 (13.94)
    FE-HS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS |  |  |  |  | 40.4 (13.4) |  |  |  | 40.4 (13.39)
    SD-CP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    SD-CP |  |  |  |  | 58.8 (15.7) |  |  |  | 58.8 (15.69)
    SD-UP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 6
    SD-UP |  |  |  |  | 39.8 (10.3) |  |  |  | 39.8 (10.26)
    MD-CP: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
    MD-CP | 63.0 (NA) — SD cannot be calculated |  |  | 46.0 (2.8) |  |  |  |  | 51.7 (10.02)
    MD-UP: number analyzed (Participants) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 6
    MD-UP | 74.5 (4.9) | 41.8 (6.9) |  |  |  |  |  |  | 52.7 (17.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This study consisted of 7 segments: 1) single ascending dose in healthy subjects (SAD-HS), 2) multiple ascending dose in healthy subjects (MAD-HS), 3) food effect in healthy subjects (FE-HS), 4) single dose in subjects with cholestatic pruritus (SD-CP), 5) multiple dose in subjects with cholestatic pruritus (MD-CP), 6) single dose in subjects with uremic pruritus (SD-UP), and 7) multiple dose in subjects with uremic pruritus (MD-UP).
  Participants
    SAD-HS: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS: Female | 8 |  | 4 |  | 5 | 4 | 3 | 1 | 25
    SAD-HS: Male | 2 |  | 2 |  | 1 | 2 | 3 | 5 | 15
    MAD-HS: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS: Female | 1 |  | 3 |  | 2 | 1 |  |  | 7
    MAD-HS: Male | 5 |  | 3 |  | 4 | 5 |  |  | 17
    FE-HS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS: Female |  |  |  |  | 3 |  |  |  | 3
    FE-HS: Male |  |  |  |  | 2 |  |  |  | 2
    SD-CP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    SD-CP: Female |  |  |  |  | 3 |  |  |  | 3
    SD-CP: Male |  |  |  |  | 2 |  |  |  | 2
    SD-UP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 6
    SD-UP: Female |  |  |  |  | 2 |  |  |  | 2
    SD-UP: Male |  |  |  |  | 4 |  |  |  | 4
    MD-CP: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
    MD-CP: Female | 1 |  |  | 1 |  |  |  |  | 2
    MD-CP: Male | 0 |  |  | 1 |  |  |  |  | 1
    MD-UP: number analyzed (Participants) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 6
    MD-UP: Female | 1 | 1 |  |  |  |  |  |  | 2
    MD-UP: Male | 1 | 3 |  |  |  |  |  |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This study consisted of 7 segments: 1) single ascending dose in healthy subjects (SAD-HS), 2) multiple ascending dose in healthy subjects (MAD-HS), 3) food effect in healthy subjects (FE-HS), 4) single dose in subjects with cholestatic pruritus (SD-CP), 5) multiple dose in subjects with cholestatic pruritus (MD-CP), 6) single dose in subjects with uremic pruritus (SD-UP), and 7) multiple dose in subjects with uremic pruritus (MD-UP).
  Participants
    SAD-HS: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS: Hispanic or Latino | 3 |  | 0 |  | 0 | 3 | 2 | 1 | 9
    SAD-HS: Not Hispanic or Latino | 7 |  | 6 |  | 6 | 3 | 3 | 4 | 29
    SAD-HS: Unknown or Not Reported | 0 |  | 0 |  | 0 | 0 | 1 | 1 | 2
    MAD-HS: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS: Hispanic or Latino | 0 |  | 0 |  | 0 | 1 |  |  | 1
    MAD-HS: Not Hispanic or Latino | 6 |  | 6 |  | 5 | 5 |  |  | 22
    MAD-HS: Unknown or Not Reported | 0 |  | 0 |  | 1 | 0 |  |  | 1
    FE-HS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS: Hispanic or Latino |  |  |  |  | 0 |  |  |  | 0
    FE-HS: Not Hispanic or Latino |  |  |  |  | 5 |  |  |  | 5
    FE-HS: Unknown or Not Reported |  |  |  |  | 0 |  |  |  | 0
    SD-CP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    SD-CP: Hispanic or Latino |  |  |  |  | 0 |  |  |  | 0
    SD-CP: Not Hispanic or Latino |  |  |  |  | 5 |  |  |  | 5
    SD-CP: Unknown or Not Reported |  |  |  |  | 0 |  |  |  | 0
    SD-UP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 6
    SD-UP: Hispanic or Latino |  |  |  |  | 0 |  |  |  | 0
    SD-UP: Not Hispanic or Latino |  |  |  |  | 6 |  |  |  | 6
    SD-UP: Unknown or Not Reported |  |  |  |  | 0 |  |  |  | 0
    MD-CP: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
    MD-CP: Hispanic or Latino | 0 |  |  | 0 |  |  |  |  | 0
    MD-CP: Not Hispanic or Latino | 1 |  |  | 1 |  |  |  |  | 2
    MD-CP: Unknown or Not Reported | 0 |  |  | 1 |  |  |  |  | 1
    MD-UP: number analyzed (Participants) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 6
    MD-UP: Hispanic or Latino | 0 | 0 |  |  |  |  |  |  | 0
    MD-UP: Not Hispanic or Latino | 2 | 4 |  |  |  |  |  |  | 6
    MD-UP: Unknown or Not Reported | 0 | 0 |  |  |  |  |  |  | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Population: This study consisted of 7 segments: 1) single ascending dose in healthy subjects (SAD-HS), 2) multiple ascending dose in healthy subjects (MAD-HS), 3) food effect in healthy subjects (FE-HS), 4) single dose in subjects with cholestatic pruritus (SD-CP), 5) multiple dose in subjects with cholestatic pruritus (MD-CP), 6) single dose in subjects with uremic pruritus (SD-UP), and 7) multiple dose in subjects with uremic pruritus (MD-UP).
  Participants
    SAD-HS Asian: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS Asian | 2 |  | 0 |  | 2 | 1 | 1 | 0 | 6
    SAD-HS Black or African American: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS Black or African American | 0 |  | 0 |  | 0 | 0 | 0 | 0 | 0
    SAD-HS White: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS White | 5 |  | 6 |  | 5 | 3 | 2 | 4 | 25
    SAD-HS American Indian or Alaska Native: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS American Indian or Alaska Native | 1 |  | 0 |  | 0 | 0 | 0 | 0 | 1
    SAD-HS Native Hawaiian or Pacific Islander: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS Native Hawaiian or Pacific Islander | 0 |  | 0 |  | 0 | 0 | 2 | 0 | 2
    SAD-HS Other: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6 | 40
    SAD-HS Other | 2 |  | 0 |  | 1 | 2 | 1 | 2 | 8
    MAD-HS Asian: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS Asian | 2 |  | 0 |  | 1 | 2 |  |  | 5
    MAD-HS Black or African American: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS Black or African American | 0 |  | 0 |  | 0 | 0 |  |  | 0
    MAD-HS White: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS White | 3 |  | 4 |  | 3 | 2 |  |  | 12
    MAD-HS American Indian or Alaska Native: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS American Indian or Alaska Native | 0 |  | 0 |  | 0 | 0 |  |  | 0
    MAD-HS Native Hawaiian or Pacific Islander: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS Native Hawaiian or Pacific Islander | 1 |  | 1 |  | 0 | 2 |  |  | 4
    MAD-HS Other: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0 | 24
    MAD-HS Other | 0 |  | 1 |  | 2 | 1 |  |  | 4
    FE-HS Asian: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS Asian |  |  |  |  | 0 |  |  |  | 0
    FE-HS Black or African American: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS Black or African American |  |  |  |  | 0 |  |  |  | 0
    FE-HS White: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS White |  |  |  |  | 5 |  |  |  | 5
    FE-HS American Indian or Native American: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS American Indian or Native American |  |  |  |  | 0 |  |  |  | 0
    FE-HS Native Hawaiian or Pacific Islander: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS Native Hawaiian or Pacific Islander |  |  |  |  | 0 |  |  |  | 0
    FE-HS Other: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
    FE-HS Other |  |  |  |  | 0 |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: To assess safety and tolerability of EP547 following single and multiple oral administration
Time Frame: Measured from Day 1 to End of Study or Early Termination (up to 3 weeks)
Population: All safety analyses were based on the Safety Population, which included all subjects who received at least one dose of study drug (EP547 or placebo).
Measure: Number; unit: participants
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Number analyzed (Participants) | 19 | 4 | 12 | 2 | 28 | 12 | 6 | 6
participants
  SAD-HS : Any TEAE: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6
  SAD-HS : Any TEAE | 5 |  | 5 |  | 5 | 3 | 3 | 4
  SAD-HS : Any Serious TEAE: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6
  SAD-HS : Any Serious TEAE | 0 |  | 0 |  | 0 | 0 | 0 | 0
  SAD-HS : Any drug-related TEAE: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6
  SAD-HS : Any drug-related TEAE | 0 |  | 2 |  | 1 | 0 | 1 | 2
  SAD-HS : Any TEAE leading to discontinuation of study drug: number analyzed (Participants) | 10 | 0 | 6 | 0 | 6 | 6 | 6 | 6
  SAD-HS : Any TEAE leading to discontinuation of study drug | 0 |  | 0 |  | 0 | 0 | 0 | 0
  MAD-HS : Any TEAE: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0
  MAD-HS : Any TEAE | 3 |  | 6 |  | 4 | 4 |  |
  MAD-HS : Any Serious TEAE: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0
  MAD-HS : Any Serious TEAE | 0 |  | 0 |  | 0 | 0 |  |
  MAD-HS : Any drug-related TEAE: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0
  MAD-HS : Any drug-related TEAE | 2 |  | 5 |  | 3 | 2 |  |
  MAD-HS : Any TEAE leading to discontinuation of study drug: number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 0 | 0
  MAD-HS : Any TEAE leading to discontinuation of study drug | 0 |  | 0 |  | 0 | 0 |  |
  FE-HS : Any TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  FE-HS : Any TEAE |  |  |  |  | 3 |  |  |
  FE-HS : Any Serious TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  FE-HS : Any Serious TEAE |  |  |  |  | 0 |  |  |
  FE-HS : Any drug-related TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  FE-HS : Any drug-related TEAE |  |  |  |  | 1 |  |  |
  FE-HS : Any TEAE leading to discontinuation of study drug: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  FE-HS : Any TEAE leading to discontinuation of study drug |  |  |  |  | 0 |  |  |
  SD-CP : Any TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  SD-CP : Any TEAE |  |  |  |  | 4 |  |  |
  SD-CP : Any Serious TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  SD-CP : Any Serious TEAE |  |  |  |  | 0 |  |  |
  SD-CP : Any drug-related TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  SD-CP : Any drug-related TEAE |  |  |  |  | 0 |  |  |
  SD-CP : Any TEAE leading to discontinuation of study drug: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  SD-CP : Any TEAE leading to discontinuation of study drug |  |  |  |  | 0 |  |  |
  SD-UP : Any TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
  SD-UP : Any TEAE |  |  |  |  | 1 |  |  |
  SD-UP : Any Serious TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
  SD-UP : Any Serious TEAE |  |  |  |  | 0 |  |  |
  SD-UP : Any drug-related TEAE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
  SD-UP : Any drug-related TEAE |  |  |  |  | 0 |  |  |
  SD-UP : Any TEAE leading to discontinuation of study drug: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
  SD-UP : Any TEAE leading to discontinuation of study drug |  |  |  |  | 0 |  |  |
  MD-CP : Any TEAE: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  MD-CP : Any TEAE | 1 |  |  | 1 |  |  |  |
  MD-CP : Any Serious TEAE: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  MD-CP : Any Serious TEAE | 0 |  |  | 0 |  |  |  |
  MD-CP : Any drug-related TEAE: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  MD-CP : Any drug-related TEAE | 0 |  |  | 1 |  |  |  |
  MD-CP : Any TEAE leading to discontinuation of study drug: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  MD-CP : Any TEAE leading to discontinuation of study drug | 0 |  |  | 0 |  |  |  |
  MD-UP : Any TEAE: number analyzed (Participants) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  MD-UP : Any TEAE | 1 | 2 |  |  |  |  |  |
  MD-UP : Any Serious TEAE: number analyzed (Participants) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  MD-UP : Any Serious TEAE | 0 | 0 |  |  |  |  |  |
  MD-UP : Any drug-related TEAE: number analyzed (Participants) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  MD-UP : Any drug-related TEAE | 0 | 0 |  |  |  |  |  |
  MD-UP : Any TEAE leading to discontinuation of study drug: number analyzed (Participants) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  MD-UP : Any TEAE leading to discontinuation of study drug | 0 | 0 |  |  |  |  |  |

2. Secondary Outcome: Maximum Plasma Concentration [Cmax] After Single Dose of EP547
Description: To evaluate the pharmacokinetics of single dose of EP547
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 9, and 12 hours post-dose on Day 1
Population: All PK analyses were based on the PK Population. For non-FE segments, the PK Population included all subjects who received ≥1 dose of EP547 and for whom a sufficient number of samples were available to determine at least 1 PK parameter.
  For FE segment, the PK Population included all randomized subjects who received ≥1 dose of EP547, had no protocol deviations affecting the PK variables of EP547, and for whom a sufficient number of samples were available to determine at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Number analyzed (Participants) | 0 | 4 | 12 | 2 | 28 | 12 | 6 | 6
ng/mL
  SAD-HS: number analyzed (Participants) | 0 | 0 | 6 | 0 | 6 | 6 | 6 | 6
  SAD-HS |  |  | 1421.0 (29.4) |  | 6309.6 (19.3) | 17232.6 (17.6) | 27799.2 (29.8) | 36352.2 (38.3)
  MAD-HS: number analyzed (Participants) | 0 | 0 | 6 | 0 | 6 | 6 | 0 | 0
  MAD-HS |  |  | 1506.6 (38.4) |  | 3973.4 (35.5) | 16954.8 (35.0) |  |
  FE-HS (Fasted): number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
  FE-HS (Fasted) |  |  |  |  | 5780.3 (22.9) |  |  |
  FE-HS (Fed): number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  FE-HS (Fed) |  |  |  |  | 3504.0 (30.0) |  |  |
  SD-CP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  SD-CP |  |  |  |  | 5019.5 (31.7) |  |  |
  SD-UP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
  SD-UP |  |  |  |  | 3483.3 (75.0) |  |  |
  MD-CP: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  MD-CP |  |  |  | 1728.5 (93.7) |  |  |  |
  MD-UP: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  MD-UP |  | 781.0 (54.6) |  |  |  |  |  |

3. Secondary Outcome: Maximum Plasma Concentration [Cmax] After Multiple Doses of EP547
Description: To evaluate the pharmacokinetics of multiple doses of EP547
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, and 24 hours post-dose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | EP547 20 mg | EP547 25 mg | EP547 30 mg | EP547 75 mg | EP547 225 mg | EP547 450 mg | EP547 675 mg
Number analyzed (Participants) | 0 | 4 | 6 | 2 | 6 | 6 | 0 | 0
ng/mL
  SAD-HS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MAD-HS: number analyzed (Participants) | 0 | 0 | 6 | 0 | 6 | 6 | 0 | 0
  MAD-HS |  |  | 2834.7 (16.4) |  | 8760.7 (27.4) | 29613.1 (21.0) |  |
  FE-HS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SD-CP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SD-UP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MD-CP: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  MD-CP |  |  |  | 3421.0 (27.8) |  |  |  |
  MD-UP: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  MD-UP |  | 3192.7 (49.5) |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Measured from Day 1 to End of Study or Early Termination (up to 3 weeks)
Description: Adverse events reporting based on the Safety Population, which included all subjects who received at least one dose of study drug (EP547 or placebo). All AE summaries restricted to treatment-emergent adverse events only.
Groups:
- SAD-HS Placebo; MAD-HS Placebo: Participants in all segments received placebo matched to EP547.
- MD-CP Placebo; MD-UP Placebo: Participants in this segment received placebo matched to EP547.
- MD-UP EP547 20 mg: Participants in this segment received 20 mg of EP547 QD for 7 days.
- SAD-HS EP547 25 mg: Participants in this segment received a single 25 mg dose of EP547.
- MAD-HS EP547 25 mg: Participants in this segment received 25 mg of EP547 QD for 7 days.
- MD-CP EP547 30 mg: Participants in this segment received 30 mg of EP547 QD for 7 days.
- SAD-HS EP547 75 mg; SD-CP EP547 75 mg; SD-UP EP547 75 mg: Participants in this segment received a single 75 mg dose of EP547.
- MAD-HS EP547 75 mg: Participants in this segment received 75 mg of EP547 QD for 7 days.
- FE-HS EP547 75 mg: Participants in this segment received a single 75 mg dose of EP547 under fed or fasted condition, separated by a washout period.
- SAD-HS EP547 225 mg: Participants in this segment received a single 225 mg dose of EP547.
- MAD-HS EP547 225 mg: Participants in this segment received 225 mg of EP547 QD for 7 days.
- SAD-HS EP547 450 mg: Participants in this segment received a single 450 mg dose of EP547.
- SAD-HS EP547 675 mg: Participants in this segment received a single 675 mg dose of EP547.
Arm/Group | SAD-HS Placebo | MAD-HS Placebo | MD-CP Placebo | MD-UP Placebo | MD-UP EP547 20 mg | SAD-HS EP547 25 mg | MAD-HS EP547 25 mg | MD-CP EP547 30 mg | SAD-HS EP547 75 mg | MAD-HS EP547 75 mg | FE-HS EP547 75 mg | SD-CP EP547 75 mg | SD-UP EP547 75 mg | SAD-HS EP547 225 mg | MAD-HS EP547 225 mg | SAD-HS EP547 450 mg | SAD-HS EP547 675 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/1 | 0/2 | 0/4 | 0/6 | 0/6 | 0/2 | 0/6 | 0/6 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/1 | 0/2 | 0/4 | 0/6 | 0/6 | 0/2 | 0/6 | 0/6 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/10 | 3/6 | 1/1 | 1/2 | 2/4 | 4/6 | 6/6 | 1/2 | 5/6 | 4/6 | 3/5 | 4/5 | 1/6 | 3/6 | 4/6 | 3/6 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD-HS Placebo (N=10) | MAD-HS Placebo (N=6) | MD-CP Placebo (N=1) | MD-UP Placebo (N=2) | MD-UP EP547 20 mg (N=4) | SAD-HS EP547 25 mg (N=6) | MAD-HS EP547 25 mg (N=6) | MD-CP EP547 30 mg (N=2) | SAD-HS EP547 75 mg (N=6) | MAD-HS EP547 75 mg (N=6) | FE-HS EP547 75 mg (N=5) | SD-CP EP547 75 mg (N=5) | SD-UP EP547 75 mg (N=6) | SAD-HS EP547 225 mg (N=6) | MAD-HS EP547 225 mg (N=6) | SAD-HS EP547 450 mg (N=6) | SAD-HS EP547 675 mg (N=6)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid skin dryness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site dermatitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site laceration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT04510090/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT04510090/SAP_001.pdf